CLINICAL TRIAL: NCT05982392
Title: Effect of Preoperative Tramadol and Naproxen Sodium on Efficacy of Local Anesthesia and Post-operative Pain in Patients With Symptomatic Irreversible Pulpitis
Brief Title: Effect of Preoperative Tramadol and Naproxen Sodium on Post Operative Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Tayyaba Tahira, Lecturer, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2889
Record Dates: First submitted 2023-07-19; First posted 2023-08-08 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Symptomatic Irreversible Pulpitis; Post Operative Pain
Keywords: Tramadol; Naproxen Sodium; Placebo
MeSH Terms: conditions — Pain, Postoperative | interventions — Tramadol; Naproxen

STUDY DESIGN:
Intervention Model Description: The participants will be randomly divided into 3 groups by envelope method. Group A will receive premedication of Oral tramadol 100mg, Group B will receive premedication of oral naproxen sodium 550mg. Both medicines will be given 60 minutes prior to the local anesthesia administration. The third group, Group C, will be the control group and no active preoperative medication will be given to these participants. A placebo will be given to these participants. These medications will be given as a single intervention only.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Clinician and participants both will be blind to the medicine given to the participants. Participants will be allowed to pick envelopes and a paramedical staff will be trained in giving medication to the participants. Procedure will be performed by an intern (who is not part of the research)Investigator will also be masked to the treatment being provided Outcome Assessor will be an intern who is not on research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tramadol (Active Comparator): Group A will receive premedication of Oral tramadol 100mg,
  Interventions: Drug: Tramadol
- Naproxen Sodium (Active Comparator): Group B will receive premedication of oral naproxen sodium 550mg.
  Interventions: Drug: Naproxen Sodium
- Placebo (Placebo Comparator): Group C, will be the control group and no active preoperative medication will be given to these patients.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tramadol — Tramadol 100mg will be given 60 minutes before start of procedure.
  Other Names: Tramal tablet
  Arms: Tramadol
Drug: Naproxen Sodium — Naproxen sodium 550mg will be given 60 minutes before start of procedure.
  Other Names: Synflex 550mg
  Arms: Naproxen Sodium
Drug: Placebo — Placebo will be given 60 minutes before start of procedure.
  Other Names: Surbex Z
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to compare in Tramadol, Naproxen sodium and Placebo in participants presenting with irreversible pulpitis in their mandibular posterior teeth.

The main question[s] it aims to answer are:

* Local anesthetic efficacy and .
* Postoperative pain. Participants will receive premedication treatments 60 minutes prior to the local anesthesia administration.

Researchers will compare Tramadol, Naproxen sodium and Placebo to evaluate their effects on Inferior alveolar nerve block efficacy and Postoperative pain.

DETAILED DESCRIPTION:
The adult participants who report in out-patient department (OPD) of Operative Dentistry at Dow International Dental College with the symptoms of irreversible pulpitis will be screened for the participation in the study. A detailed history will be taken which will be followed by clinical examination and complemented with sensibility testing with Endo Ice or electric pulp test. Radiographic analysis will also be done to confirm the diagnosis to assess for factors pertaining to exclusion and inclusion criteria. Verbal and written informed consent will be taken from all the participants.

Randomization: The participants will be randomly divided into 3 groups by envelope method.

Group A will receive premedication of Oral tramadol 100mg, Group B will receive premedication of oral naproxen 550mg. Both medicines will be given 60 minutes prior to the local anesthesia administration. The third group, Group C, will be the control group and no active preoperative medication will be given to these participants. A placebo will be given to these participants. These medications will be given as a single intervention only.

Blinding: Clinician and participants both will be blind to the medicine given to the participants. Participants will be allowed to pick envelopes and a paramedical staff will be trained in giving medication to the participants.

Pain scores will be recorded by asking the participant to rate their pain on a scale ranging from 0 to 10 before medication and then after 15 minutes, 30 minutes and 60 minutes of administering the premedication. Pain score will also be recorded after 10 minutes of the administration of Inferior alveolar nerve block (IANBs) and buccal nerve block & during deroofing process of chamber opening.

Two cartridges of Lidocaine 1.8 ml having a concentration of 1:100,000 of Epinephrine will be used for administration of regional anesthesia. Access opening will be performed under rubber dam isolation with a Mani number 245 bur in a high-speed hand piece with copious water irrigation. Sodium hypochlorite (5.25%) will be used as a standard root canal irrigation solution.Pulpectomy will be performed with Mani K-files (8-25) till respective working lengths of the teeth under study.

To assess the post-operative pain, a proforma and pain intensity scale will be provided to the participants for self recording at 6, 24, 48 and 72 hours after the procedure. The participants will return the proforma to an intern on 3rd day to be assessed by an intern supervised by the principal investigator.

(For this research, "The investigators will be offering As per need analgesic for breakthrough pain. Participants will be offered brufen 400mg as needed. The participants will be advised to mark breakthrough pain on VAS at the time of taking medicine).

The participants will also be monitored for the adverse effects of these medications (nausea, vomiting, dizziness, drowsiness) as a secondary outcome .at above-mentioned time-intervals.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and ASA II individuals who are between the ages of 18 and 60 years.
* Patients who have been diagnosed with symptomatic irreversible pulpitis (with either a normal periapex or symptomatic apical periodontitis).
* Patients who score moderate to severe (4-10) on a preoperative visual analogue scale (VAS= 1-10).
* Mandibular permanent premolar and molars.

Exclusion Criteria:

* Patients who had taken painkillers or narcotics in the previous 12 hours
* Patients suffering from severe pain because of traumatic occlusion.
* Teeth with extensive damage, calcified canals, root resorption, and an open apex.
* Previously root canal treated teeth.
* Medically compromised patients (ASA-III and above)
* Those with special communication needs or who do not understand Urdu or English language.
* Pregnant and lactating women
* Individual patients who will be driving back alone
* Patients who are allergic to the prescribed medicines

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Local Anesthesia Efficacy | 10minutes,20minutes
  Change in pain will be assessed after administration of inferior alveolar nerve block and during access opening on a visual analogue scale of 0-10 ," 0 being no pain", "10 being worst pain"
Postoperative pain | 6 hours, 24 hours,48 hours, 72hours
  Change in pain will be assessed after cleaning and shaping till #25 k file on a visual analogue scale of 0-10, "0 being no pain and 10 being worst pain"

SECONDARY OUTCOMES:
Adverse effects of Medications | 6hours, 24hours
  Nausea, Headache, Dizziness, Vertigo will be recorded as experienced or not experienced

CONTACTS AND LOCATIONS:
Overall Officials: Tayyaba Tahira, BDS FCPS, Principal Investigator — Dow International Dental College, Dow University of Health Sciences; Farah Naz, BDS FCPS, Study Director — Dow International Dental College, Dow University of Health Sciences
Locations (1):
- Dow International Dental College, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Only investigators and co-investigators of this study will be able to access to participants' personal data.
  Ownership of the data will remain with the principal investigator and Department of Operative Dentistry, Dow International Dental College